CLINICAL TRIAL: NCT02762006
Title: A Phase Ib Trial of Neoadjuvant Durvalumab (MEDI4736) +/- Tremelimumab in Locally Advanced Renal Cell Carcinoma
Brief Title: Neoadjuvant MEDI 4736 +/- Tremelimumab in Locally Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moshe Ornstein (Other)
Responsible Party: Sponsor-Investigator, Moshe Ornstein, MD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12815
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: durvalumab; tremelimumab; Phase Ib; Locally Advanced
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab with Nephrectomy (Experimental): Following systemic therapy, patients will undergo nephrectomy. Adjuvant therapy will be administered within 4-6 weeks of surgery. Subsequent follow-up will then be completed to assess adverse event resolution and long-term outcomes.
  * Cohort 1: Durvalumab x 1 dose (n=6)
  * Cohort 2: Durvalumab + Tremelimumab x 1 dose (n=6)
  * Cohort 2a: Durvalumab + Tremelimumab x 1 dose (n=12)
  * Cohort 3: Durvalumab + Tremelimumab x 1 dose (n=9)
  Cohorts 1 and 2: Adjuvant dosing of Durvalumab x 1 beginning 2-8 weeks after surgery.
  Cohort 2a: Durvalumab monotherapy until 1 year after nephrectomy.
  Cohort 3: Adjuvant dosing of durvalumab + tremelimumab x 1 beginning 2-8 weeks after surgery, then durvalumab monotherapy until 1 year after nephrectomy.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a programmed cell death ligand-1 monoclonal antibody which has demonstrated anti-tumor efficacy renal cell carcinoma and other malignancies via activation of the immune system.
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab is a CTLA-4 monoclonal antibody.

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of administering investigational drugs (meaning not Food and Drug Administration (FDA)-approved for kidney cancer) prior to surgical treatment for kidney cancer. The first drug is called MEDI4736, and the second drug is called tremelimumab. Both of these drugs work by attaching to certain proteins on immune cells with the goal of stimulating an immune response against cancer cells. This is a phase 1 trial, with the primary goal of identifying if this treatment is safe and possible side effects when given prior to surgery for kidney cancer.

DETAILED DESCRIPTION:
Objectives:

Primary Objective

• To investigate the safety and feasibility of neoadjuvant plus adjuvant dosing of durvalumab +/- tremelimumab in patients with localized renal cell carcinoma (RCC).

Secondary Objectives

* To assess the immune response to neoadjuvant plus adjuvant dosing of durvalumab +/- tremelimumab in patients with localized RCC as measured an increased density of tumor-infiltrating CD8 T-cells.
* To assess the antitumor effect of neoadjuvant durvalumab +/- tremelimumab in patients with RCC as measured by change in tumor size.

Correlative Objectives

* To explore pharmacodynamic and microbiome markers of response to checkpoint inhibition in pre- and post-treatment blood and tissue samples (e.g. infiltration of T cells, T regulatory cells and/or Myeloid-derived suppressor cells).
* To understand changes in the immunological milieu mediated by pre-surgical immune checkpoint blockade (e.g. change in T cell repertoire, expression of T cell agonist targets).

Study Design:

This study will be a single-arm open-label phase Ib study of neoadjuvant durvalumab +/- tremelimumab in localized / locally advanced, non-metastatic RCC patients suitable for nephrectomy. Upon selection as appropriate for study, patients will undergo computed tomography (CT)-guided biopsy of renal mass to obtain histological confirmation of diagnosis, and immunologic characterization of the RCC tumor. Peripheral blood will also be drawn at time of screening. Patients will subsequently receive systemic neoadjuvant treatment in one of 5 cohorts as defined below. Following systemic therapy, patients will undergo nephrectomy. Type of surgery (open vs. minimally invasive, radical vs. partial) and template for lymph node dissection are at the discretion of surgeon. Timing of surgery in relation to adverse events and/or treatment for adverse events from neoadjuvant dosing of study drugs is at the discretion of the surgeon. Adjuvant therapy will be administered within 4-6 weeks of surgery. Subsequent follow-up will then be completed to assess adverse event resolution and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of renal cell carcinoma (any histologic subtype) without evidence of distant metastatic disease
* Patients must have clinical stage T2b-4 and/or N1, M0 disease
* Written informed consent and any locally-required authorization (e.g., HIPAA)) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate normal organ and marrow function as defined below:

  * Hemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (≥ 1500 per mm3)
  * Platelet count ≥ 100 x 109/L (≥100,000 per mm3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with the study sponsor.
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
  * Glomerular filtration rate > 40ml/min/1.73m2 as estimated by the Cockcroft-Gault formula or creatinine clearance >50ml/min as determined by 24-hour urine collection:
  * Estimated creatinine clearance (Clcr) in mL/min by the Cockcroft-Gault (C-G): {[140 - age ( years)]× weight (kg)}/{72 × serum creatinine (mg / dL)} ×0.85 for female patients
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study.
* Participation in another clinical study with an investigational product during the last 30 days.
* Prior systemic anti-cancer therapy of any kind for RCC, including but not limited to any approved agent or any previous treatment with a PD1 or PD-L1 inhibitor including durvalumab. No previous treatment with immunotherapy for any malignancy including cytokine, anti-tumor vaccine, T-cell activator, co-stimulator or immune checkpoint inhibitor.
* Evidence of metastatic renal cell carcinoma on imaging and/or biopsy. Involvement of regional lymph nodes is permitted.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from an electrocardiogram (ECG) using Fridericia's Correction (QTcF).

  * a. At Screening, a single ECG will be obtained on which QTcF must be <470 ms. In case of clinically significant ECG abnormalities, including a QTcF value >470 ms, 2 additional 12-lead ECGs should be obtained over a brief period (eg, 30 minutes) to confirm the finding.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Active or prior documented autoimmune disease within the past 2 years.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to tremelimumab or any excipient
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension (defined as >160/90 mmHg despite medical therapy), unstable angina pectoris (requiring nitrates), cardiac arrhythmia (NOT including controlled atrial fibrillation), active peptic ulcer disease or gastritis, active bleeding diathesis including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C (detectable RNA) or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control

  * Pregnant or breastfeeding women are excluded from this study.
* Subjects with uncontrolled seizures
* Subjects with known HIV, active hepatitis B, or active hepatitis C (detectable RNA). HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with durvalumab and/or tremelimumab. In addition, these subjects are at increased risk of lethal infections when treated with immunosuppressive therapy.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Patients with Dose Limiting Toxicity (DTL) | Up to 12 months after screening
  Dose-limiting toxicities (DLTs) will be evaluated from the first dose of drug through the first adjuvant dose of durvalumab. Grading of DLTs will follow the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Average estimated blood loss during nephrectomy | Up to 56 days after screening
Average operative time (hours) | Up to 56 days after screening
Average length of hospital stay (days) | Up to 56 days after screening
Average days in the intensive care unit (ICU) | Up to 56 days after screening
Average volume of post operative blood transfusion | Up to 56 days after screening
Number of patients with perioperative complications by grade of the Clavien-Dindo Classification System | Up to 56 days after screening
  * Grade 1
    * Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions
    * Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics, electrolytes, and physiotherapy. This grade also includes wound infections opened at the bedside
  * Grade II
    -- Requiring pharmacological treatment with drugs other than such allowed for grade I complications
  * Blood transfusions and total parenteral nutrition are also included
    --Grade III - Requiring surgical, endoscopic or radiological intervention
  * Grade IIIa - Intervention not under general anesthesia
  * Grade IIIb - Intervention under anesthesia
  * Grade IV - Life-threatening complication (including CNS complications) requiring IC/ICU management
  * Grade IVa - Single organ dysfunction (including dialysis)
  * Grade IVb - Multiorgan dysfunction
  * Grade V - Death of a patients
Percentage of tumor-infiltrating CD8+ T-cells after treatment | Up to 12 months after screening
  The primary readout here will be increased CD8 infiltration versus a large historical control cohort already in our possession. Preliminary studies will focus on peri-tumoral and inter-tumoral CD8 infiltration, as those parameters are associated with responsiveness to immunotherapy in melanoma patients. Secondary efforts will focus on the induction of a pro-inflammatory infiltrate by comparing the surgical specimen to pre-treatment biopsies. Those assays will be challenged by the small amount of tissue generally available from biopsy, but are important since the biopsy could potentially serve as a valuable prediction tool to guide early treatment.
Tumor response rate according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 12 months after screening
  RECIST 1.1 Criteria Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Proportion of patients with measurable disease according to RECIST 1.1 | Up to 12 months after screening
Best overall response rate (BOR) according to RECIST 1.1 | Up to 12 months after screening
  o The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ornstein, MD, MA, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio